CLINICAL TRIAL: NCT05864170
Title: the Safety and Efficacy Evaluation of HGI-001 Injection in Patients With Transfusion-Dependent β-Thalassemia(Child)
Brief Title: the Safety and Efficacy Evaluation of HGI-001 Injection in Patients With Transfusion-Dependent β-Thalassemia
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Shenzhen Hemogen (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HGI-001-CTP
Record Dates: First submitted 2023-02-28; First posted 2023-05-18 (Actual); Last update posted 2024-11-29 (Actual); Status verified 2024-11

CONDITIONS: β-thalassemia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental (Experimental): Three transfusion-dependent β-thalassaemia subjects aged 18-35 years will be reinfused with β-globin restored autologous hematopoietic stem cells modified with LentiHBBT87Q
  Interventions: Biological: β-globin restored autologous hematopoietic stem cells

INTERVENTIONS:
Biological: β-globin restored autologous hematopoietic stem cells — β-globin-restored autologous hematopoietic stem cells modified with LentiHBBT87Q

SUMMARY:
This is an open label study to evaluate the safety and efficacy of β-globin Restored Autologous Hematopoietic Stem Cells in ß-Thalassemia Major Patients

DETAILED DESCRIPTION:
We will recruit ß-thalassaemia major patients and collect their autologous hematopoietic stem cells, which will be modified with the LentiHBBT87Q system to restore β-globin expression. After conditioning, the autologous hematopoietic stem cells with restored β-globin will be reinfused to the patients and followed up for two years to collect data.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 18-35 years (inclusive), ICF can be provided by the patient and/or legal guardian;
2. Definitively diagnosed with severe TDT without genotype restriction, and a valid test report can be provided;
3. Average transfusion volume > 100 mL/kg/year or transfusion frequency > 8 times/year within 2 years prior to enrollment, or has been definitively diagnosed with TDT;
4. At least 3 months of full volume transfusion (verification of blood transfusion records can be provided) prior to screening, and Hb is maintained at ≥ 9.0 g/dL;
5. Ferritin load < 3000 μg/L, cardiac and liver iron indicates moderate or lesser iron overload; records of iron chelation treatments within 3 months before screening (including prescription or receipt) can be provided;
6. Acceptable organ functions (including heart, liver, kidney, lung and coagulation functions), stable disease condition, and suitable for busulfan pre-treatment and hematopoietic stem cell (HSC) transplantation as judged by the investigator;
7. Meets follow-up requirements, adheres to treatment arrangements, and is able to return to the hospital regularly to undergo various examinations within 2 years after reinfusion of HGI-001 injection.

Exclusion Criteria:

1. Patients with fully HLA-matched donors;
2. Received allogeneic transplantation, which needs to be weighed and evaluated by an expert committee; received other gene therapies;
3. Have previously undergone splenectomy;
4. Uncorrected bleeding disorder;
5. Uncontrolled epilepsy and mental illness;
6. Received hydroxyurea, ruxolitinib, decitabine, or cytarabine within 3 months prior to enrollment;
7. Psychoactive substance abuse, drug or alcohol abuse within 6 months prior to enrollment;
8. Patients with pulmonary hypertension who have not been given effective intervention;
9. Persistent toxicity (≥ CTCAE grade 2) induced by previous treatment;
10. Positive for anti-RBC antibodies in antibody screening;
11. Positive for hepatitis B surface antigen (HBsAg) and HBV DNA copy number > upper limit of normal (ULN) (HBV DNA test not required for patients negative for HBsAg), positive for hepatitis C virus (HCV) antibody, positive human immunodeficiency virus (HIV), or positive for Treponema pallidum antibody (TP-Ab) (subjects who are positive for the antibody due to vaccination can be enrolled). In certain clinical environments/regions, subjects who are positive for other tests can also be excluded from the trial, such as, human lymphocytic virus-1 (HTLV-1) or -2 (HTLV-2), tuberculosis, and toxoplasmosis.
12. Has or has had malignant tumors or myeloproliferative disease or immunodeficiency disease;
13. Immediate family member with or suspected of having a familial cancer (including but not limited to hereditary breast and ovarian cancers, nonpolyposis colorectal cancer, and adenomatous polyposis);
14. Severe bacterial, viral, fungal or parasitic infection;
15. Other illnesses which render the subject unsuitable for participation (e.g., severe liver, kidney or heart disease); Definition of severe liver and kidney disease: a. Aspartate aminotransferase (AST), alanine aminotransferase (ALT), or total bilirubin > 3 × ULN; b. Liver magnetic resonance imaging (MRI) indicates significant cirrhosis; c. Liver biopsy indicates cirrhosis, severe fibrosis or active hepatitis (liver biopsy is only performed when liver MRI indicates active hepatitis and significant fibrosis without evidence for cirrhosis); d. Creatinine clearance < 30% of normal;
16. WBC < 3 × 109/L and/or PLT < 100 × 109/L;
17. Has diabetes, abnormal thyroid functions or other endocrine disorder;
18. Participated in other interventional clinical studies within 4 weeks before the trial;
19. Poor adherence or other conditions that renders the subject unsuitable for participation as judged by the investigator.

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 3 (Estimated)
Dates: Start 2022-05-27 (Actual); Primary Completion 2025-12-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Overall response rate | 24 months
  Percent of patients with average VCN > 0.1 in peripheral blood mononuclear cells (PBMCs) and average expression of exogenous adult hemoglobin HbAT87Q > 2.0 g/dL
Incidence and severity of AEs | 0-24 months
  The number and the percentage of adverse events related to transplantation will be summarized according to NCI CTCAE 5.0
Incidence of SAEs | 0-24 months
  The number of SAE related to transplantation will be summarized according to NCI CTCAE 5.0
Transplantation-related fatal and disabling events within day 100 after transplantation | Day 100
  Transplantation-related fatal and disabling events
Overall survival rate during the clinical trial | 0-24 months
  Number of patients alive through the whole trial will be record
HGI-001 injection-related replicating lentivirus test | 0-24 months
  The percentage of RCL should be negative in the 24 months after transplant
Change from baseline in Clonal variations containing specific viral integration sites | 0-24 months
  Evaluation of the percentage of participants without abnormal clonal proliferation and polyclonal engraftment at 6, 12, 18 and 24 months after transplant. More than 1000 VIS retrieved from peripheral blood should be checked.
Number of patients with abnormal hematology and bone marrow cytology within 24 months after reinfusion, and percent of patients with abnormal RBC proliferation | 0-24 months
  Number of patients with abnormal hematology and bone marrow cytology

SECONDARY OUTCOMES:
Treatment response rate | 12 Months
  Percent of patients with average VCN > 0.1 in PBMCs and average expression of exogenous adult hemoglobin HbAT87Q > 2.0 g/dL after reinfusion of HGI-001 injection
Percent of subjects with successful HSC engraftment | 1 month
  Criteria for successful engraftment: Absolute neutrophil count > 0.5 × 10 9 /L for 3 consecutive days; platelet count is maintained at > 20 × 10 9 /L for 7 consecutive days without platelet transfusion
Change in transfusion volume or frequency | 0-24 Months
  Change in average annual transfusion volume or frequency from baseline or change in percentage
Transfusion improvement rate | 0-24 Months
  Percent of subjects with ≥ 30% decrease in the average annual (0-12 months, 12-24 months) transfusion volume or frequency from baseline after reinfusion of HGI-001 injection
Transfusion independence (TI) rate | 0-24 Months
  Percent of subjects who do not require transfusion for at least 12 consecutive months after reinfusion of HGI-001 injection and have a weighted average Hb of ≥ 9.0 g/dL
Transfusion-free survival | 0-24 Months
  the time when a subject meets the TI criteria and maintains transfusion-free survival
Changes in VCN and exogenous adult HbAT87Q expression | 0-24 Months
  Vector copy number
Changes in cardiac iron load after reinfusion of HGI-001 injection | 0-24 Months
  T2 MRI
Changes in liver iron load after reinfusion of HGI-001 injection | 0-24 Months
  T2 MRI
Changes in serum ferritin after reinfusion of HGI-001 injection | 0-24 Months
  serum ferritin
Changes use of iron chelation medications after reinfusion of HGI-001 injection | 0-24 Months
  iron chelation medications

CONTACTS AND LOCATIONS:
Overall Officials: Chao Liu, PHD, Principal Investigator — Shenzhen Hemogen; Li Yu, Principal Investigator — Shenzhen University General Hospital
Locations (1):
- Shenzhen University General Hospital, Shenzhen, Guangdong, China